CLINICAL TRIAL: NCT06737757
Title: Prospective, Multicenter, Randomized Controlled, Non-Inferiority Clinical Trial Evaluating the Safety and Efficacy of Artificial Polymer Heart Valve for the Treatment of Aortic Valve Disease
Brief Title: Clinical Trial Evaluating the Safety and Efficacy of Artificial Polymer Heart Valve for the Treatment of Aortic Valve Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suzhou Hearthill Medical Technology Co.,LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PoliaValve-SA-02
Record Dates: First submitted 2024-12-11; First posted 2024-12-17 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Aortic Valve Stenosis; Aortic Valve Disease; Aortic Valve Regurgitation
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve Disease; Aortic Valve Insufficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group(PoliaValve) (Experimental): Using artificial polymer heart valves(PoliaValve, Hearthill Medical) for aortic valve replacement
  Interventions: Device: Artificial polymer heart valves
- Control Group (Active Comparator): Using bovine pericardium aortic valve for aortic valve replacement
  Interventions: Device: Bovine pericardial aortic valve

INTERVENTIONS:
Device: Artificial polymer heart valves — The experimental group will use polymer material surgical aortic valves(PoliaValve, Hearthill Medical) for aortic valve replacement
  Arms: Experimental group(PoliaValve)
Device: Bovine pericardial aortic valve — The control group will undergo aortic valve replacement using bovine pericardial aortic valve
  Arms: Control Group

SUMMARY:
The purpose of this study is to conduct the clinical investigation of the HeartHill Medical's polymer aortic valve, namely PoliaVavle，to collect evidence on the device's safety and performance. This prospective, multicenter, randomized controlled, non inferiority clinical trial is expected to enroll 198 subjects and conduct a 1:1 random grouping. The experimental group will use polymer material surgical aortic valves（PoliaVavle, HeartHill Medical, Suzhou China) for aortic valve replacement, while the control group will use bovine pericardial biological valves for aortic valve replacement.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects are aged ≥18 years old;
2. The subjects understand the nature and purpose of the study, voluntarily participate, and sign the informed consent form. They agree to comply with the trial requirements, cooperate with surgical treatment and follow-up, and consent to relevant follow-up inquiries and examinations;
3. The subjects have been confirmed to have severe aortic valve stenosis and/or regurgitation (also known as insufficiency) through echocardiography;
4. According to the 2020 ACC/AHA guidelines for the management of patients with valvular heart disease, the subjects meet the indications for surgical aortic valve replacement and preoperative assessment recommends surgical aortic valve replacement.

Exclusion Criteria:

1. Other valve diseases with surgical indications, such as severe mitral regurgitation, severe tricuspid regurgitation, moderate or greater mitral stenosis, or a history of previous aortic or other valve replacement surgery;
2. Other severe cardiovascular conditions with surgical indications, such as Stanford A-type aortic dissection, aortic sinus aneurysm (sinus diameter > 5.0cm), hypertrophic obstructive cardiomyopathy, diffuse three-vessel coronary artery disease, or placement of a left ventricular assist device in end-stage heart failure;
3. End-stage heart failure that is not reversible even with aortic valve surgery, such as severe left ventricular dysfunction (LVEF < 25%), or severe heart failure that cannot be corrected, or severe pulmonary hypertension assessed by right heart catheterization, with planned postoperative Impella, IABP, or left ventricular assist;
4. Preoperative decompensated heart failure, cardiogenic shock, malignant arrhythmias, etc., requiring mechanical circulatory support, mechanical ventilation, or emergency surgery;
5. Active endocarditis within the past 3 months or the presence of cardiac vegetations;
6. Severe acute myocardial infarction or history of cerebrovascular accidents within the past 3 months (excluding lacunar infarcts);
7. Severe renal insufficiency (glomerular filtration rate < 30mL/min) or end-stage renal disease requiring long-term dialysis;
8. Liver dysfunction or gastrointestinal malnutrition-related diseases;
9. Active bleeding, bleeding tendencies, or patients unable to receive anticoagulant therapy;
10. Severe respiratory or ventilatory dysfunction requiring continuous oxygen therapy;
11. Poor compliance or cognitive impairment (such as coma, Parkinson's disease, dementia, substance abuse), inability to follow study requirements or refusal to participate in follow-up visits;
12. Other conditions with an expected lifespan of less than 1 year, such as malignancies and immunodeficiency diseases;
13. Other situations not suitable for artificial aortic valve replacement or participation in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Survival rate without prosthetic valve events at 12 months post-surgery | 12 months following patient enrollment completion
  Event-free survival of the prosthetic valve at 12 months postoperatively. The 12-month postoperative survival rate without artificial valve events. The event-free survival rate refers to patients who have not experienced any reasons for heart-related or non-heart-related deaths, moderate or severe artificial valve degeneration, or the need for re-intervention on the artificial valve within 12 months after surgery.

SECONDARY OUTCOMES:
Surgical success rate | 1 month following patient enrollment completion
  Surgical success rate: Surgical success is defined as the prosthetic valve function within 1 month after surgery, the prosthetic valve has a transvalvular pressure difference of <20mmHg or a peak flow rate of < 3m/s, no moderate or above intravalvular regurgitation or paravalvular leakage), and the patient survives without re-intervention.
Evaluation of postoperative artificial valve function(effective valve orifice area) | baseline and 12months following patient enrollment completion
  Use echocardiography to evaluate the effective valve orifice area to assess the hemodynamic Performance.
Evaluation of postoperative artificial valve function(mean transvalvular pressure gradient) | baseline and 12months following patient enrollment completion
  Use echocardiography to evaluate the mean transvalvular pressure gradient.
Evaluation of postoperative artificial valve function(peak flow velocity) | baseline and 12months following patient enrollment completion
  Use echocardiography to measure the peak flow velocity.
Evaluation of postoperative artificial valve function(regurgitation) | baseline and 12months following patient enrollment completion
  Evaluate the presence or absence of intravalvular or paravalvular regurgitation during the follow-up period by echocardiography.
New York Heart Association Assessment (NYHA) | baseline and 12months following patient enrollment completion
  Evaluate the New York Heart Association (NYHA) assessment to determine the improvement in cardiac function.The NYHA classification of heart function consists of four levels, ranging from Class I to Class IV, with heart function progressively deteriorating.
Left ventricular ejection fraction(LVEF) change from baseline in postoperative echocardiographic | baseline and 12 months post-surgery
  LVEF(%) change from baseline in postoperative echocardiography.
Left ventricular end-systolic diameter(LVESD) change from baseline in postoperative echocardiographic | baseline and 12 months post-surgery
  LVESD(mm) change from baseline in postoperative echocardiography.
Left ventricular end-diastolic diameter(LVEDD) change from baseline in postoperative echocardiographic | baseline and 12 months post-surgery
  LVEDD(mm) change from baseline in postoperative echocardiography.
BNP or NT-proBNP | baseline and 12 months following patient enrollment completion
  Measure BNP or NT-proBNP to get the changes in postoperative cardiac function from baseline.

OTHER OUTCOMES:
The incidence of device-related adverse events | 12months following patient enrollment completion
  The incidence of device-related adverse events: Valve-related complications include moderate or greater structural valve degeneration, valve thrombosis, valve-related thromboembolism, severe bleeding (due to anticoagulant use), severe paravalvular leak, and prosthetic valve endocarditis.
Surgical adverse event rate | 12months following patient enrollment completion
  Surgical adverse event rate: Surgical complications include severe lung infections, mediastinal or incision infections, postoperative severe hypotension, perioperative stroke, new-onset atrial fibrillation, new-onset complete atrioventricular block, acute kidney injury or worsening renal function requiring renal replacement therapy, severe bleeding, and cardiac tamponade.
Incidence of structural valve degeneration | 12months following patient enrollment completion
  Incidence of structural valve degeneration: Structural valve degeneration refers to valve stenosis and/or regurgitation due to structural abnormalities of the valve itself (such as tearing, shedding, calcification, fibrosis, deformation of the valve frame, and rupture of the connecting parts between the valve components) as determined by reoperation or clinical examination (e.g., echocardiography, etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Fanglin Lu, MD, Study Chair — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine; Xiangbin Pan, MD, Study Chair — Chinese Academy of Medical Sciences, Fuwai Hospital